CLINICAL TRIAL: NCT03152838
Title: The Role of Epigenetic Modifications in Autism Spectrum Disorder Through DNA Methylation
Brief Title: The Role of Epigenetic Modifications in Autism Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Mohammed Ali, principal investigator, Assiut University
Other Study IDs: HRM
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Cases: 20 confirmed autism cases will be involved in this study.
  1. The autism patients will be diagnosed according to:Gilliam Autism Rating Scale Arabic version: An assessment of the severity of autism using the Gilliam autism rating scale Arabic version: This test was used for diagnosis and assessment of the severity of autistic features for ages 3-22 years. It consists of 56 items, subdivided into 4 subscales: communication, social interaction, stereotyped behaviors, development and total score.
  2. Fasting blood samples will be collected from autism children for DNA Methylation-and quantitative Real-time Polymerase Chain Reaction Analysis
  Interventions: Genetic: DNA methylation and Real-time Polymerase Chain Reaction Analysis; Diagnostic Test: Gilliam Autism Rating Scale Arabic version
- Control: 20 age-gender matched typical development children that will be assigned to the normal control group.
  1. Control children will be examined by a psychiatrist to exclude any sub-clinical autistic features.
  2. Fasting blood samples will be collected from control children for DNA Methylation-and quantitative Real-time Polymerase Chain Reaction Analysis
  Interventions: Genetic: DNA methylation and Real-time Polymerase Chain Reaction Analysis

INTERVENTIONS:
Genetic: DNA methylation and Real-time Polymerase Chain Reaction Analysis — Fasting blood samples will be collected from both autism and controls for DNA extraction. Peripheral blood (2ml) will be drawn from the cubital vein intoplastic syringes. Lymphocytes will be isolated from blood samples. We will examine the gene methylation in the peripheral blood lymphocytes of drug-naı¨ve autism patients and control subjects.
  DNA will be isolated from lymphocytes, purified and processed for bisulfate modification. Bisulfate treatment of genomic DNA will be performed using DNA methylation kit according to the manufacturer´ instructions. Bisulfite treatment of genomic DNA converts cytosine to uracil, but leaves methylated 5'Cytosines unchanged. Quantitative real time Polymerase chain reaction will be used to determine the DNA methylation status of the Brian derived neurotrophic factor and glia fibrillary acidic protein genes using primers specific to the human genes.
Diagnostic Test: Gilliam Autism Rating Scale Arabic version — An assessment of the severity of autism using the Gilliam autism rating scale Arabic version: This test was used for diagnosis and assessment of the severity of autistic features for ages 3-22 years. It consists of 56 items, subdivided into 4 subscales: communication, social interaction, stereotyped behaviors, development and total score. The Arabic version has been validated with good reliability and validity and used in many studies before. The lower the scores are, the worse the condition is.
  The scale will be done by trained and certified psychologist. The protocol and informed consent for this study will be reviewed and approved by the ethics committee at the Faculty of Medicine, Assiut University, Egypt.
  Groups: Autism Cases

SUMMARY:
Autism Spectrum Disorder is a neurodevelopmental disorder characterized by impaired social communication and repetitive or stereotyped behaviors. According to the World Health Organization , the prevalence of Autism Spectrum Disorder is one person in 160.

DETAILED DESCRIPTION:
Genetic and non-genetic factors would contribute to the development of autism. However, the molecular mechanisms of ASD are not clear and successful treatments are still under research. Autism Spectrum Disorder can occur due to exposure to environmental pollutants which lead to epigenetic changes like DNA methylation, acetylation and post-translational modifications. However, the role of epigenetic changes in Autism Spectrum Disorder is still debated.

Epigenetic mechanisms represent a link through which environmental factors interact with the genetic factors resulting in modification of Autism Spectrum Disorder risk through changes in gene expression. DNA methylation and histone deacetylation are two major epigenetic mechanisms that regulate the gene expression at successive stages of brain development.

Brain derived neurotrophic factor is responsible for brain development. Altered BDNF levels and expression may be closely associated with Autism Spectrum Disorder. . Glial fibrillary acidic protein is the hallmark intermediate filament protein in astrocytes, the main type of glial cells in the central nervous system. Interestingly, Glial fibrillary acidic protein is a marker of astroglial activation and the recent data indicated that Glial fibrillary acidic protein could be implicated in the pathophysiology of autism. However, the underlying mechanisms for the role of brain derived neurotrophic factor and glial fibrillary acidic protein in autism spectrum disorder are poorly understood.

ELIGIBILITY:
Inclusion Criteria:

1. - All enrolled children with Autism Spectrum Disorder will be:

   1. Exhibit symptoms within the typical triad of autistic traits: communication impairment, social deficits, and ritualistic interests.
   2. Drug-naïve.
2. Children with Autism Spectrum Disorder and controls will be 2-6 years old.

Exclusion Criteria:

The control subjects will also clinically examined by the psychiatrist to exclude any sub-clinical autistic features. Children with Autism Spectrum Disorder and controls will excluded from the study if

1. They receive treatment for any reason.
2. -Endocrinological disease, mental retardation, communication disorder, psychotic disorder, attention deficit hyperactivity disorder and learning disorders seen in the children or their family members.

Ages: 2 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: The children attending the pediatric clinic at Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
The difference of percentage of DNA methylation of Brain derived neurotrophic factor gene and glial fibrillary acidic protein gene between the two groups | one year
  Real Time Polymerase Chain Reaction
The relation between the severity of autistic symptoms and percentage of Brain derived neurotrophic factor gene and glial fibrillary acidic protein gene methylation in Autism cases group | one year
  correlation test

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bahi A. Sustained lentiviral-mediated overexpression of microRNA124a in the dentate gyrus exacerbates anxiety- and autism-like behaviors associated with neonatal isolation in rats. Behav Brain Res. 2016 Sep 15;311:298-308. doi: 10.1016/j.bbr.2016.05.033. Epub 2016 May 17. PMID 27211062
- [Result] Bhandari R, Kuhad A. Resveratrol suppresses neuroinflammation in the experimental paradigm of autism spectrum disorders. Neurochem Int. 2017 Feb;103:8-23. doi: 10.1016/j.neuint.2016.12.012. Epub 2016 Dec 23. PMID 28025035
- [Result] Gladkevich A, Kauffman HF, Korf J. Lymphocytes as a neural probe: potential for studying psychiatric disorders. Prog Neuropsychopharmacol Biol Psychiatry. 2004 May;28(3):559-76. doi: 10.1016/j.pnpbp.2004.01.009. PMID 15093964
- [Result] Paternain L, Martisova E, Campion J, Martinez JA, Ramirez MJ, Milagro FI. Methyl donor supplementation in rats reverses the deleterious effect of maternal separation on depression-like behaviour. Behav Brain Res. 2016 Feb 15;299:51-8. doi: 10.1016/j.bbr.2015.11.031. Epub 2015 Nov 25. PMID 26628207
- [Result] Vuong HE, Hsiao EY. Emerging Roles for the Gut Microbiome in Autism Spectrum Disorder. Biol Psychiatry. 2017 Mar 1;81(5):411-423. doi: 10.1016/j.biopsych.2016.08.024. Epub 2016 Aug 26. PMID 27773355
- [Result] Wang J, Zou Q, Han R, Li Y, Wang Y. Serum levels of Glial fibrillary acidic protein in Chinese children with autism spectrum disorders. Int J Dev Neurosci. 2017 Apr;57:41-45. doi: 10.1016/j.ijdevneu.2017.01.004. Epub 2017 Jan 11. PMID 28088366
- [Result] Nishimura K, Nakamura K, Anitha A, Yamada K, Tsujii M, Iwayama Y, Hattori E, Toyota T, Takei N, Miyachi T, Iwata Y, Suzuki K, Matsuzaki H, Kawai M, Sekine Y, Tsuchiya K, Sugihara G, Suda S, Ouchi Y, Sugiyama T, Yoshikawa T, Mori N. Genetic analyses of the brain-derived neurotrophic factor (BDNF) gene in autism. Biochem Biophys Res Commun. 2007 Apr 27;356(1):200-6. doi: 10.1016/j.bbrc.2007.02.135. Epub 2007 Mar 5. PMID 17349978
- [Result] Ferreira MC, Dorboz I, Rodriguez D, Boespflug Tanguy O. Screening for GFAP rearrangements in a cohort of Alexander disease and undetermined leukoencephalopathy patients. Eur J Med Genet. 2015 Sep;58(9):466-70. doi: 10.1016/j.ejmg.2015.07.002. Epub 2015 Jul 21. PMID 26208460
- [Result] Samadi SA, McConkey R. The utility of the Gilliam autism rating scale for identifying Iranian children with autism. Disabil Rehabil. 2014;36(6):452-6. doi: 10.3109/09638288.2013.797514. Epub 2013 Jun 5. PMID 23738615